## Title: Standardized Patients to Measure and Address Intersectional Stigma

Date: September 12, 2022

Clinicaltrial.gov Identifier: NCT04896216

Version: 1.6

## **Provider Consent Form**

Study title: STD and Sexual Health Clinic Diagnosis and Treatment Service Research

Hello! You have been invited to participate in a research project run by the University of Minnesota and the Guangdong Provincial Dermatology Hospital. The purpose of this project is to learn about work environments and training opportunities for dermatovenerology providers in Guangzhou. The ultimate goal of this study is to create and evaluate professional skills building workshop to help providers like you improve patient-centered care in facilities like yours. By patient-centered care we are referring to care based on values such as respect for patients' preferences or provision of education and information.

What will I need to do to participate? Today, we will ask you to fill out a short survey about yourself and your medical training, the services offered at this institution, and your clinical experience. We estimate that this survey will take approximately 15 minutes to complete. Later, at sometime within the next 6 months, we will send a trained member of our survey team to visit your office, posing as a regular patient. S/He will not identify themselves to you at that time, and you may think s/he is just another patient. If you suspect that someone you are treating is a fake patient, we ask that you do not confront him/her during the visit and rather simply continue to treat him/her as you would any other patient. If you'd like, you can write down the patient's name and a description; at the end of the study you will have an opportunity to check with us as to whether or not someone was a fake patient. We estimate that the time you spend with the "fake patient" will be no more than 30 minutes. Afterwards, the SP will record what happened during the visit using a standard checklist. This information will be used for research purposes only. No one outside of the research team will have access to this information, including you, your colleagues, or your supervisors. Our goal in using these fake patients is to design a better training program for providers like you and to evaluate its effectiveness.

About a year after these fake patient visits we will invite you to a hybrid professional skills building workshop at the Guangdong Center for STD Control & Prevention. With the consideration of the pandemic and your work schedule, we provide a hybrid workshop to minimize the travel and gathering, which includes online pre-workshop videos, and attending the in-person training (42 dollars / 300 RMB compensation for each participant). Participation in the workshop is voluntary, and all workshop related costs including travel and accommodations will be covered by the study.

Starting about one month after the workshop and then over the next six months, fake patients will once more conduct unannounced clinic visits using the same data collection techniques described previously.

Lastly about a year after the workshop our study staff will conduct a final visit with you to readminister a similar survey as we will complete today. At that point in time you can check with us about any suspected fake patient visits.

There will be no cost to you for any of the study activities or procedures.

**Will being in this study help me in any way?** There are no direct benefits to you as a participant for taking part in this study. However, views and experiences that you share with us throughout the study will help us better understand your work environment and the healthcare services available to your patients. It may also help us design a more optimal training workshop

for providers like you, which could benefit you if local policy makers choose to roll out this type of training.

Is there any way that being in this study could be bad for me? Some survey questions may be difficult to answer, and you do not have to answer any question that makes you feel uncomfortable. If you experience any discomfort while answering questions you should report any problems to the researcher. In addition, there is a small risk that of a breach of data security for information about you or your facility, which could expose your providers to scrutiny about the quality of healthcare provided here. To minimize this risk all data collection procedures with the fake patients will take place inside vehicles rented for the purpose of visiting facilities (vehicle drivers will be asked to step outside of the vehicle during data collection). At the soonest convenience all study materials and data related to your facility or providers will be replaced with codes, and its linkages to any identifying information will be accessible only to the study leadership and senior staff.

What happens to the information collected for this research? Only study leaders and team members with proper training in research ethics and data security will have access to information that identifies you. These will be the only individuals permitted to analyze and interpret the data. All documents and files related to your facility or providers will be stored on encrypted and password protected tablets or computers stored at our secured study office. All personally identifying information collected about you will be destroyed once it is no longer needed for the study. No presentation or publication of the study results will refer to participants individually. Manuscripts published regarding this work will be based on the de-identified database. Finally, any breaches of confidentiality or unanticipated problems that occur during the study will be brought to attention of the two study leaders, Drs. Kumi Smith and Sean Sylvia, who will notify the IRBs of the University of Minnesota and GDCDC for further review and action.

What happens if I say "yes" but change my mind later? At any time and for any reasons you may quit this study without any penalty. If you have an unexpected reaction or fail to follow the instructions, the investigator also has the right to stop your participation. Should you choose to withdraw, our study staff will offer you a choice between having whatever existing data we have collected from you retained or discarded. Please be aware that even if you withdraw, information about the facility where you work or from some of your colleagues will likely still make it into the final analysis.

What if later I think of other questions I have about this study? If you have any questions, complaints or concerns, please contact Dr. Wang Cheng, Director of the STD Control Department at the Guangdong Provincial Dermatology Hospital at (20) 87255824 and GDDH@protonmail.com. You should also contact him at any time if you feel you have been hurt by being a part of this study, if you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant.

By completing this survey, you are giving your consent to be in this study.